CLINICAL TRIAL: NCT07297602
Title: Evaluation of Efficacy and Safety of Oral Roflumilast in Treatment of Moderate to Severe Atopic Dermatitis: a Pilot Study
Brief Title: Evaluation of Efficacy and Safety of Oral Roflumilast for Treatment of Moderate to Severe Atopic Dermatitis in Patients Aged 12 Years and Older: A Pilot Study
Acronym: ROFLU-AD12
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nora Mohamed Abdelrazik (Other)
Collaborators: Mansoura University Hospital (Other)
Responsible Party: Sponsor-Investigator, Nora Mohamed Abdelrazik, Lecturer of Dermatology, Mansoura University Hospital
Organization: Mansoura University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R.25.11.3442.R1
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; Oral roflumilast; Moderate-to-severe AD; Efficacy; Safety; Adolescents and Adults
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Roflumilast; Tablets

STUDY DESIGN:
Intervention Model Description: This is a single-arm, open-label pilot study in which all participants, both male and female, receive oral roflumilast. Participants will not be randomized to different treatments. Male and female participants will be analyzed as subgroups to explore potential sex-based differences in safety and efficacy. No placebo or comparator group is included.
Masking Description: This is an open-label study: neither the participants nor the investigators are blinded. All participants receive oral roflumilast, and both participants and study staff are aware of the treatment assignment. No placebo or comparator is used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation of Oral Roflumilast in Moderate to Severe Atopic Dermatitis (Experimental): All participants, both male and female, will receive oral roflumilast. No placebo or comparator is included. Male and female participants will be analyzed as subgroups for exploratory safety and efficacy outcomes.
  Interventions: Drug: Oral roflumilast

INTERVENTIONS:
Drug: Oral roflumilast — Participants will receive oral roflumilast. The initial dose is 250 mcg once daily for the first 10 days, followed by a dose escalation to 500 mcg once daily for the remainder of the 12-week treatment period.
  Route: Oral Schedule: Daily for 12 weeks Duration: 12 weeks
  Other Names: Roflumilast (generic name); Daxas (brand name in some countries); Roflumilast 500 mcg tablet (formulation identifier)

SUMMARY:
This is a 12-week, single-arm, open-label pilot study to assess the safety and preliminary efficacy of oral roflumilast in patients aged 12 years and older with moderate-to-severe atopic dermatitis All participants, both male and female, will receive oral roflumilast starting at 250 mcg once daily for 10 days, followed by 500 mcg once daily for the remainder of the study. The primary outcome is the mean change in SCORAD (Scoring Atopic Dermatitis) score from baseline to Week 12. Secondary outcome include safety assessments, including treatment-emergent adverse events, serious adverse events, and laboratory abnormalities. Male and female participants will be analyzed as subgroups to explore potential differences in response or safety.

ELIGIBILITY:
Inclusion Criteria:

* AD patients ≥ 12 years in whom systemic therapy is indicated.
* Patients who don't use other systemic therapy for AD in the last 2 months (or naïve who didn't use any systemic therapy before).
* Safe contraception during the study.

Exclusion Criteria:

* Pregnant or lactating women, as well as women of childbearing potential not using an effective method of contraception.
* Age <12 years.
* Other concomitant AD systemic treatments such as cyclosporins and biologics.
* Previous systemic treatment of AD in the last 2 months.
* Patients receiving inducers or inhibitors of cytochromes CYP3A4 and CYP1A.
* Other systemic diseases other than COPD, especially hepatic impairment.
* Hypersensitivity to the active substance of roflumilast or to any of its excipients.
* The use of contraception with gestodene and ethinylestradiol.
* Unreliable patients.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-05-20 (Estimated)

PRIMARY OUTCOMES:
The primary outcome of the study is the change in the SCORAD Index from baseline to the end of treatment | Baseline and Weeks 4, 8, and 12.
  SCORAD is a validated scoring system that provides a comprehensive assessment of atopic dermatitis by combining:
  Extent of eczema: The percentage of total body surface area affected (0-100%), assessed using standard dermatologic mapping.
  Intensity of clinical signs: Six features-erythema, swelling ,oozing/crusts, scratch marks, lichenification, and dryness-each graded from 0 (absent) to 3 (severe).
  Patient-reported symptoms: Daily pruritus (itch) and sleep disturbance, each rated on a 0-10 visual analogue scale.
  The total SCORAD score ranges from 0 to 103, with higher values indicating more severe disease.
  Changes in SCORAD are reported as:
  Absolute reduction, and
  Percentage improvement from baseline (e.g., SCORAD-50 or SCORAD-75).
  This outcome measure captures both objective clinical improvement and patient-experienced symptom relief, providing a holistic evaluation of treatment efficacy.

SECONDARY OUTCOMES:
Safety - incidence of treatment-emergent adverse events and laboratory abnormalities. | Throughout treatment; labs at baseline and monthly (Weeks 4, 8, 12).
  Incidence and severity of adverse events (including diarrhea, nausea, abdominal pain, weight loss, decreased appetite, insomnia, headache) and clinically significant changes in CBC, hepatic profile, and serum creatinine.

CONTACTS AND LOCATIONS:
Overall Officials: Abeer Mohamed Elkholy, MD Dermatology, Study Chair — Faculty of medicine, Mansoura University
Locations (1):
- Mansoura University Hospital, Al Mansurah, Dakahlia Governorate, Egypt